CLINICAL TRIAL: NCT01966471
Title: A Randomized, Multicenter, Open-Label, Phase III Trial Comparing Trastuzumab Plus Pertuzumab Plus a Taxane Following Anthracyclines Versus Trastuzumab Emtansine Plus Pertuzumab Following Anthracyclines as Adjuvant Therapy in Patients With Operable HER2-Positive Primary Breast Cancer
Brief Title: A Study of Trastuzumab Emtansine (Kadcyla) Plus Pertuzumab (Perjeta) Following Anthracyclines in Comparison With Trastuzumab (Herceptin) Plus Pertuzumab and a Taxane Following Anthracyclines as Adjuvant Therapy in Participants With Operable HER2-Positive Primary Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO28407; 2012-004902-82 (EudraCT Number)
Record Dates: First submitted 2013-10-17; First posted 2013-10-21 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; Trastuzumab; pertuzumab; Paclitaxel; Epirubicin; Doxorubicin; Docetaxel; Cyclophosphamide; Fluorouracil

ARMS (2):
- Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane (Active Comparator): Trastuzumab and pertuzumab will be administered concurrently for up to a total duration of 1 year (up to 18 cycles [1 Cycle = 21 days]) with the taxane (docetaxel or paclitaxel) component of chemotherapy following anthracycline [5 fluorouracil, epirubicin, and cyclophosphamide (FEC) or epirubicin and cyclophosphamide (EC) or doxorubicin and cyclophosphamide (AC)] based chemotherapy.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Drug: Epirubicin; Drug: Doxorubicin; Drug: Docetaxel; Drug: Cyclophosphamide; Drug: 5-Fluorouracil
- Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab (Experimental): Trastuzumab emtansine and pertuzumab will continue for up to a total duration of 1 year (up to 18 cycles [1 Cycle = 21 days]) following anthracycline [5 fluorouracil, epirubicin, and cyclophosphamide (FEC) or epirubicin and cyclophosphamide (EC) or doxorubicin and cyclophosphamide (AC)] based chemotherapy.
  Interventions: Drug: Trastuzumab Emtansine; Drug: Epirubicin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Trastuzumab Emtansine — Trastuzumab emtansine IV infusion (duration 90 minutes) will be administered at 3.6 mg/kg q3w for up to 18 cycles (1 cycle = 21 days).
  Other Names: Kadcyla
  Arms: Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Drug: Trastuzumab — Trastuzumab IV infusion (duration 90 minutes) will be administered at 8 mg/kg loading dose followed by 6 mg/kg IV q3w for up to 18 cycles (1 cycle = 21 days).
  Other Names: Herceptin
  Arms: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane
Drug: Pertuzumab — Pertuzumab infusion (duration 60 minutes) will be administered at 840 mg loading dose followed by 420 mg IV q3w for up to 18 cycles (1 cycle = 21 days).
  Other Names: Perjeta
  Arms: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane
Drug: Paclitaxel — IV infusion of paclitaxel 80 mg/m^2 once weekly may be administered concurrently with trastuzumab in combination with pertuzumab for 12 weeks.
  Arms: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane
Drug: Epirubicin — 3 to 4 cycles (1 cycle = 21 days) of standard of care anthracycline-based chemotherapy using epirubicin may be administered in both Arms 1 and 2 as per discretion of the investigator and local prescribing information/institutional guidelines.
Drug: Doxorubicin — 3 to 4 cycles (1 cycle = 21 days) of standard of care anthracycline-based chemotherapy using doxorubicin may be administered in both Arms 1 and 2 as per discretion of the investigator and local prescribing information/institutional guidelines.
Drug: Docetaxel — IV infusion either docetaxel every 3 weeks (q3w) (at 100 milligram per square meter [mg/m^2] for 3 cycles (1 cycle = 21 days); at 75 mg/m2 for 4 cycles; or start at 75 mg/m^2 in the first cycle and escalate to 100 mg/m^2 if no dose limiting toxicity occurs, for a total of 3 cycles at minimum) may be administered concurrently with trastuzumab in combination with pertuzumab.
  Arms: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane
Drug: Cyclophosphamide — 3 to 4 cycles (1 cycle = 21 days) of standard of care anthracycline-based chemotherapy using cyclophosphamide (FEC) may be administered in both Arms 1 and 2 as per discretion of the investigator and local prescribing information/institutional guidelines.
Drug: 5-Fluorouracil — 3 to 4 cycles (1 cycle = 21 days) of standard of care anthracycline-based chemotherapy using 5-fluorouracil, may be administered in both Arms 1 and 2 as per discretion of the investigator and local prescribing information/institutional guidelines.

SUMMARY:
This two-arm, randomized, open-label, multicenter study will evaluate the efficacy and safety of trastuzumab emtansine in combination with pertuzumab versus trastuzumab in combination with pertuzumab and a taxane as adjuvant therapy in participants with human epidermal growth (HER) factor 2 (HER2)-positive primary invasive breast cancer. Following surgery and anthracycline-based chemotherapy, participants will receive either trastuzumab emtansine at a dose of 3.6 milligrams per kilogram (mg/kg) and pertuzumab at a dose of 420 milligrams (mg) intravenously (IV) every 3 weeks (q3w) or trastuzumab at a dose of 6 mg/kg and pertuzumab at a dose of 420 mg IV q3w in combination with a taxane.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (</=) 1
* Non-metastatic histologically confirmed primary invasive breast carcinoma that was operable
* HER2-positive breast cancer
* Known hormone receptor status of the primary tumor
* Adequately excised: participants must have undergone either breast-conserving surgery or mastectomy/nipple- or skin-sparing mastectomy
* Pathological tumor-node-metastasis staging (Union for International Cancer Control-American Joint Committee on Cancer [UICC/AJCC] 7th edition): eligible participants must have either:

Node-positive disease (pN more than or equal to [>/=] 1), any tumor size except T0, and any hormonal receptor status; or Node-negative disease (pN0) with pathologic tumor size >2.0 centimeters by standard local assessment and negative for estrogen receptor (ER) and progesterone receptor (PR) determined by a central pathology laboratory

* Participants with synchronous bilateral invasive disease are eligible only if both lesions are HER2-positive
* No more than 9 weeks (63 days) may elapse between definitive breast surgery (or the last surgery if additional resection required for breast cancer) and randomization
* Baseline left ventricular ejection fraction (LVEF) >/=55% measured by echocardiogram (ECHO; preferred) or multiple-gated acquisition (MUGA) scans
* Documentation on hepatitis B virus (HBV) and hepatitis C virus (HCV) serology is required
* Female participants of childbearing potential must be willing to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception. For male participants with partners of childbearing potential, one highly effective form of contraception or two effective forms of contraception must be used. Contraception must continue for the duration of study treatment and for 6 months after the last dose of study treatment

Exclusion Criteria:

* History of any prior (ipsilateral and/or contralateral) invasive breast carcinoma
* History of non-breast malignancies within the 5 years prior to randomization, except for carcinoma in situ (CIS) of the cervix, CIS of the colon, melanoma in situ, and basal cell and squamous cell carcinomas of the skin
* Any clinical T4 tumor as defined by tumor-node-metastasis classification in UICC/AJCC 7th edition, including inflammatory breast cancer
* For the currently diagnosed breast cancer, any previous systemic anti-cancer treatment (for example, neoadjuvant or adjuvant), including but not limited to, chemotherapy, anti-HER2 therapy (for example, trastuzumab, trastuzumab emtansine, pertuzumab, lapatinib, neratinib, or other tyrosine kinase inhibitors), hormonal therapy, OR anti-cancer radiation therapy (RT) (intra-operative radiotherapy as a boost at the time of primary surgery is acceptable)
* Previous therapy with anthracyclines, taxanes, or HER2-targeted therapy for any malignancy
* History of DCIS and/or lobular CIS (LCIS) that was treated with any form of systemic chemotherapy, hormonal therapy, or RT to the ipsilateral breast where invasive cancer subsequently developed. Participants who had their DCIS/LCIS treated with surgery only and/or contralateral DCIS treated with radiation are allowed to enter the study
* Participants with contraindication to RT while adjuvant RT is clinically indicated
* Concurrent anti-cancer treatment in another investigational trial
* Cardiopulmonary dysfunction as defined by protocol: angina pectoris requiring anti-anginal medication, serious cardiac arrhythmia not controlled by adequate medication, severe conduction abnormality, or clinically significant valvular disease, significant symptoms (Grade >/=2) relating to left ventricular dysfunction, cardiac arrhythmia, or cardiac ischemia, myocardial infarction within 12 months prior to randomization, uncontrolled hypertension, evidence of transmural infarction on electrocardiogram (ECG), requirement for oxygen therapy
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness, uncontrolled infections, uncontrolled diabetes, or known infection with HIV
* Any known active liver disease. For participants who are known carriers of HBV/HCV, active hepatitis B/C infection must be ruled out per local guidelines
* Inadequate hematologic, renal or liver function
* Pregnant or lactating women
* Hypersensitivity to any of the study medications or any of the ingredients or excipients of these medications, including hypersensitivity to benzyl alcohol
* Chronic immunosuppressive therapies, including systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1846 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (295):
- United States (50):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - Kaiser Permanente - Oakland, Oakland, California
  - Kaiser Permanente - Roseville; Oncology Pharmacy, Roseville, California
  - Kaiser Permanente - Sacramento; Oncology Pharmacy, Sacramento, California
  - UC Davis Cancer Center; Oncology, Sacramento, California
  - Southern California Kaiser Permanente, San Diego, California
  - Kaiser Permanente - San Jose, San Jose, California
  - Kaiser Permanente - San Leandro, San Leandro, California
  - Kaiser Permanente - South SF; Oncology Clinical trials, South San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Kaiser Permanente - Walnut Creek; Oncology Pharmacy, Walnut Creek, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists; SCRI, Fort Myers, Florida
  - Florida Cancer Specialists; Saint Petersburg, St. Petersburg, Florida
  - University Cancer & Blood Center, LLC; Research, Athens, Georgia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Central Georgia Cancer Care PC, Macon, Georgia
  - Quincy Medical Group; Canc Ctr at Blessing Hosp, Quincy, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Anne Arundel Health System Research Instit-Annapolis Oncology Ctr, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Karmanos Cancer Institute.., Detroit, Michigan
  - Henry Ford Hospital; Hematology Oncology, Detroit, Michigan
  - US oncology research at Minnesota Oncology, Saint Paul, Minnesota
  - Mercy Medical Research Institute, Springfield, Missouri
  - Dartmouth Hitchcock Med Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - ProHEALTH Care Associates LLP, Lake Success, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Mercy Clinic Oklahoma Communties, Inc, Oklahoma City, Oklahoma
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - West Clinic, Germantown, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders - Fort Worth, Fort Worth, Texas
  - Wellmont Medical Associates, Bristol, Virginia
  - University of Virginia Health System; Hematology/Oncology Division, Charlottesville, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Blue Ridge Cancer Care - Salem, Salem, Virginia
  - University of Washington, Seattle, Washington
- Australia (8):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Calvary Mater Newcastle; Medical Oncology, Waratah, New South Wales
  - Haematology & Oncology Clinics of Australia Research Centre, South Brisbane, Queensland
  - Burnside War Memorial Hospital, Clinical Trials Centre, Adelaide, South Australia
  - Frankston Hospital; Oncology/Haematology, Frankston, Victoria
  - Austin Hospital; Medical Oncology, Heidelberg, Victoria
  - Epworth HealthCare; Clinical Trials Centre, Richmond, Victoria
  - St John of God Murdoch Hospital; Oncology West, Murdoch, Western Australia
- Belgium (2):
  - UZ Leuven Gasthuisberg, Leuven
  - Sint Augustinus Wilrijk, Apotheek, Wilrijk
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (8):
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Sirio Libanes; Centro de Oncologia, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Hospital Paulistano, São Paulo, São Paulo
- Canada (18):
  - Tom Baker Cancer Centre-Calgary, Calgary, Alberta
  - BC Cancer - Kelowna (Sindi Ahluwalia Hawkins Centre), Kelowna, British Columbia
  - Lions Gate Hospital, North Vancouver, British Columbia
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Regional health authority A vitalite health network, Moncton, New Brunswick
  - Queen Elizabeth II Health Sciences Centre; Oncology, Halifax, Nova Scotia
  - Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Credit Valley Hospital/Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Southlake Regional Health Center; Community Care Clinic / Oncology, Newmarket, Ontario
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - North York General Hospital, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Cite de La Sante de Laval; Hemato-Oncologie, Laval, Quebec
  - McGill University; Glen Site; Oncology, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- Chile (2):
  - Instituto Oncologico del sur, Temuco
  - ONCOCENTRO APYS; Oncología, Viña del Mar
- Oncomedica S.A., Montería, Colombia
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni Nemocnice Hradec Kralove; Dept of Radiotherapy & Oncology, Hradec Králové
  - MULTISCAN, s.r.o., Radiologicke centrum Pardubice, Pardubice
  - Vseobecna fakultni nemocnice v Praze, Prague
- Hospital Diagnostico Escalón, San Salvador, El Salvador
- France (24):
  - Ico - Paul Papin, Angers
  - Clinique Sainte Catherine, Avignon
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Institut Bergonie; Oncologie, Bordeaux
  - CHU de Brest - Hôpital de Morvan, Brest
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Jean Perrin; Oncologie, Clermont-Ferrand
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - Clinique Victor Hugo; Chimiotherapie, Le Mans
  - Centre Oscar Lambret; Cancerologie Gynecologique, Lille
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Centre D'Oncologie de Gentilly; Oncology, Nancy
  - Centre Antoine Lacassagne, Nice
  - Institut de cancerologie du Gard, Nîmes
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Centre Armoricain de Radiotherapie, de Imagerie Medicale et de Oncologie (CARIO), Plérin
  - Polyclinique De Courlancy; Centre Radiotherapie Oncologie, Reims
  - Centre Eugene Marquis; Service d'oncologie, Rennes
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Institut De Cancerologie De La Loire; Consult Oncologie Niveau 0, Saint-Priest-en-Jarez
  - Institut d'oncologie de l'Orangerie; Chimiotherapie, Strasbourg
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Centre Alexis Vautrin; Oncologie Medicale, Vandœuvre-lès-Nancy
- Georgia (3):
  - LTD Institute of Clinical Oncology, Tbilisi
  - Khechinashvili University Hospital ;Breast Unit, Tbilisi
  - Chemotherapy and Immunotherapy Clinic Medulla, Tbilisi
- Germany (24):
  - Klinikum Augsburg, Augsburg
  - Hochwaldkrankenhaus, Bad Nauheim
  - Frauenarzt-Zentrum Zehlendorf an der Teltower Eiche, Berlin
  - Gemeinschaftspraxis Dr. Bueckner und Dr. Nueckel, Bochum
  - Praxis Dr.med. Katja Ziegler-Löhr, Cologne
  - BAG Freiberg-Richter, Jacobasch, Illmer, Wolf; Gemeinschaftspraxis Hämatologie-Onkologie, Dresden
  - AGAPLESION Markus-Krankenhaus, Frankfurt
  - Städtische Kliniken Frankfurt am Main Höchst, Frankfurt
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Dres.Jochen Wilke und Harald Wagner, Fürth
  - Niels-Stensen-Kliniken Franziskus-Hospital Harderberg GmbH, Georgsmarienhütte
  - Universitätsklinikum Hamburg-Eppendorf; Frauenklinik, Hamburg
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Klinikum Kulmbach; Frauenklinik, Kulmbach
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Klinikum Meiningen Klinik f.Gynäkologie und Geburtshilfe, Meiningen
  - Klinikum der Universität München; Campus Großhadern; Klinik und Poliklinik für Frauenheilkunde, München
  - Hämatologisch/Onkologische Praxis Prof. Dr. Decker, Studienzentrum, Ravensburg
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Gynäkologie Kompetenzzentrum; Praxis Dr. med. Carsten Hielscher, Stralsund
  - Dres. Helmut Forstbauer, Carsten Ziske und Kollegen; Onkologische Schwerpunktpraxis, Troisdorf
  - GRN-Klinik Weinheim; Abt.Gynäkologie und Geburtshilfe, Weinheim
  - Klinikum Worms; Frauenklinik; Klinik für Gynäkologie und Geburtshilfe, Worms
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hong Kong (3):
  - Princess Margaret Hospital; Oncology, Hong Kong
  - Tuen Mun Hospital; Clinical Oncology, Hong Kong
  - Queen Mary Hospital; Dept of Surgery, Pokfulam
- Hungary (4):
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Municipal Hospital of Uzsoki Utca; Centre of Oncoradiology, Budapest
  - Debreceni Egyetem, Klinikai Kozpont, Onkologiai Klinika, Debrecen
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Israel (2):
  - Chaim Sheba Medical Center; Oncology Dept, Ramat Gan
  - Sourasky / Ichilov Hospital; Oncology Department, Tel Aviv
- Italy (15):
  - Ospedale Antonio Perrino; Oncologia Medica, Brindisi, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi; Unità Operativa Oncologia Medica, Bologna, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Policlinico Universitario Campus Biomedico; Uoc Oncologia Medica, Rome, Lazio
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - ASST DI CREMONA; Unità di Patologia Mammaria Senologia e Breast Unit, Cremona, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 1, Milan, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - Istituto Clinico Humanitas;U.O. Oncologia Medica Ed Ematologia, Rozzano, Lombardy
  - Humanitas Centro Catanese Di Oncologia; Oncologia Medica, Misterbianco (CT), Sicily
  - Ospedale Misericordia E Dolce; Oncologia Medica, Prato, Tuscany
  - Azienda Ospedaliera S. Maria - Terni; Oncologia, Terni, Umbria
  - IOV - Istituto Oncologico Veneto - IRCCS; Oncologia Medica II, Padua, Veneto
- Japan (32):
  - Aichi Cancer Center Hospital, Breast Oncology, Aichi
  - Nagoya City University Hospital; Breast Surgery, Aichi
  - Natl Hosp Org Shikoku; Cancer Ctr, Surgery, Ehime
  - National Hospital Organization Kyushu Cancer Center;Breast Oncology, Fukuoka
  - Gunma University Hospital; Department of Breast and Endocrine Surgery, Gunma
  - Gunma Prefectural Cancer Center; Breast Oncology, Gunma
  - Hiroshima City Hiroshima Citizens Hospital; Breast Surgery, Hiroshima
  - Hiroshima University Hospital; Breast Surgery, Hiroshima
  - Hyogo College Of Medicine; Breast And Endocrine Surgery, Hyōgo
  - Sagara Hospital; Breast Surgery, Kagoshima
  - St. Marianna University School of Medicine Hospital, Breast and Endocrine Surgery, Kanagawa
  - Tokai University Hospital, Breast Surgery, Kanagawa
  - Kumamoto City Hospital, Breast and Endocrine Surgery, Kumamoto
  - Kumamoto Shinto General Hospital; Breast Cancer Center, Kumamoto
  - Kyoto University Hospital; Breast Surgery, Kyoto
  - Niigata Cancer Ctr Hospital; Breast Surgery, Niigata
  - Iwate Med Univ School of Med; Surgery, Numakunai
  - Kawasaki Medical School Hospital; Breast and Thyroid Surgery, Okayama
  - Naha-nishi Clinic; Surgery, Okinawa
  - National Hospital Organization Osaka National Hospital; Breast Surgery, Osaka
  - Osaka International Cancer Institute; Breast and Endocrine Surgery, Osaka
  - Saitama Medical University International Medical Center; Breast Oncology, Saitama
  - Saitama Cancer Center, Breast Oncology, Saitama
  - Shizuoka Cancer Center; Breast Surgery, Shizuoka
  - Shizuoka General Hospital; Breast Surgery, Shizuoka
  - Jichi Medical University; Breast Oncology, Tochigi
  - National Cancer Center Hospital; Medical Oncology, Tokyo
  - St. Luke's Internat. Hospital, Breast Surgical Oncology, Tokyo
  - Tokyo Metropolitan; Komagome Hospital, Surgery, Tokyo
  - The Cancer Inst. Hosp. of JFCR; Breast Oncology Center, Tokyo
  - Showa University Hospital; Breast Surgery, Tokyo
  - Tokyo Medical Uni. Hospital; Breast Oncology, Tokyo
- Mexico (4):
  - Instituto Nacional De Cancerologia; Oncology; Tumores Mamarios, Distrito Federal
  - Fundacion Rodolfo Padilla Padilla A.C., León
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
  - Hospital San Jose Del Tec. de Monterrey; Oncology, Monterrey
- Norway (2):
  - Oslo universitetssykehus HF, Ullevål, Kreftsenteret, Oslo
  - Helse Stavanger HF, Stavanger Universitetssjukehus; Klinikk for Blod og kreftsykdommer, Stavanger
- Centro Hemato Oncologico Panama, Panama City, Panama
- Peru (4):
  - Clinica de Especialidades Medicas, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Clinica San Borja, Lima
  - Instituto Oncologico Miraflore, Miraflores
- Philippines (2):
  - San Juan de Dios Hospital;Oncology Unit, Pasay
  - East Avenue Medical Center, Quezon City
- Poland (8):
  - Bialostockie Centrum Onkologii; Oddzial Onkologii Klinicznej, Bialystok
  - Centrum Onkologii;Im. Franciszka Lukaszczyka;Onkologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kliniki Onkologii, Krakow
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii; Poradnia Chemioterapii, Lodz
  - Centrum Onkologii Ziemi LUBELSKIEJ im. Sw Jana z Dukli, I oddz. Chemioterapii, Lublin
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad; Klinika Nowtw.Piersi i Chir.Rekonstr, Warsaw
- Romania (4):
  - Institutul Oncologic Prof. Dr. Al. Trestioreanu Bucuresti, Bucharest
  - Cluj Clinical County Hospital; Oncology Dept, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - Regional Institute of Oncology Iasi, Iași
- Russia (7):
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Republican Clinical Oncologic Dispensary of Republic Of Tatarstan, Kazan'
  - FSBI Russian Oncology Research Center n.a. Blokhin of MOH RF, Moscow
  - State Inst. Of Healthcare Orenburg Regional Clinical Oncology Dis, Orenburg
  - SBI for HPE "Ryazan State Medical University n.a. I.P. Pavlov" of MoH of RF, Ryazan
  - Scientific Research Institute n.a. N.N. Petrov, Saint Petersburg
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
- Singapore (2):
  - National University Hospital; National University Cancer Institute, Singapore (NCIS), Singapore
  - National Cancer Centre; Medical Oncology, Singapore
- South Korea (5):
  - National Cancer Center; Medical Oncology, Gyeonggi-do
  - Ajou Uni Hospital; Medical Oncology, Gyeonggi-do
  - Seoul National Uni Hospital; Dept. of Internal Medicine/Hematology/Oncology, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
- Spain (11):
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Hospital de Cruces; Servicio de Oncologia, Bilbao, Vizcaya
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Centro Oncologico MD Anderson Internacional; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria; Servicio de Oncologia, Málaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (3):
  - Sahlgrenska Universitetssjukhuset; Jubileumskliniken, Gothenburg
  - Universitetssjukhuset Örebro, Onkologiska kliniken, Örebro
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (3):
  - Kantonsspital Graubünden Medizin Onkologie; Onkologie und Hämatologie, Chur
  - Luzerner Kantonsspital; Medizinische Onkologie, Lucerne
  - Brust-Zentrum Zürich AG Seefeldstrasse 214 Zürich, Zurich
- Taiwan (6):
  - Changhua Christian Hospital; Dept of Surgery, Changhua
  - Kaohsiung Medical Uni Chung-Ho Hospital; Dept of Surgery, Kaohsiung City
  - Taichung Veterans General Hospital; Dept of Surgery, Taichung
  - VETERANS GENERAL HOSPITAL; Department of General Surgery, Taipei
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Tri-Service General Hospital, Division of General Surgery, Taipei
- Thailand (4):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Chiang Rai Prachanukroh Hospital; Department Of Medicine, Chiang Rai
  - Buddhachinaraj Phitsanulok Hospital; Chemotherapy Unit ; Department of Medicine, Phitsanuok
- Ukraine (2):
  - State Medical Academy; Oncology, Dnipropetrovsk
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
- United Kingdom (22):
  - Velindre Cancer Centre; Oncology Dept, Cardiff
  - Cheltenham General Hospital; Gloucestershire Oncology Centre, Cheltenham
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Cornwall
  - University Hospital Coventry; InHANSE Unit and Clinical Trials Cancer Treatment Centre, Coventry
  - Western General Hospital; Edinburgh Breast Unit, Edinburgh
  - Royal Devon & Exeter Hospital; Oncology Centre, Exeter
  - Royal Surrey County Hospital; St. Lukes Cancer Centre, Guildford
  - Leicester Royal Infirmary; Dept. of Medical Oncology, Leicester
  - Royal Marsden Hospital - Fulham; Oncology Department, London
  - Charing Cross Hospital, London
  - Maidstone Hospital; Kent Oncology Centre, Maidstone
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - Freeman Hospital; Northern Centre For Cancer Care, New Castle Upon Tyne
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham City Hospital; Oncology, Nottingham
  - Peterborough City Hospital, Edith Cavell Campus; Oncology Department, Peterborough
  - Queen Alexandra Hospital; Portsmouth Haematology & Oncology Centre, Level B, Portsmouth
  - Weston Park Hospital; Cancer Clinical Trials Centre, Sheffield
  - Musgrove Park Hospital; Department Clinical Research, Beacon Centre, Somerset
  - Uni Hospital of North Staffordshire; Staffordshire Oncology Centre, Stoke-on-Trent
  - Royal Marsden Hospital; Dept of Medical Oncology, Sutton
  - Yeovil District Hospital; Macmillan Cancer Unit, Yeovil

REFERENCES:
- [Derived] Krop IE, Im SA, Barrios C, Bonnefoi H, Gralow J, Toi M, Ellis PA, Gianni L, Swain SM, Im YH, De Laurentiis M, Nowecki Z, Huang CS, Fehrenbacher L, Ito Y, Shah J, Boulet T, Liu H, Macharia H, Trask P, Song C, Winer EP, Harbeck N. Trastuzumab Emtansine Plus Pertuzumab Versus Taxane Plus Trastuzumab Plus Pertuzumab After Anthracycline for High-Risk Human Epidermal Growth Factor Receptor 2-Positive Early Breast Cancer: The Phase III KAITLIN Study. J Clin Oncol. 2022 Feb 10;40(5):438-448. doi: 10.1200/JCO.21.00896. Epub 2021 Dec 10. PMID 34890214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 288 centers in 36 countries.
Pre-assignment Details: Randomization was stratified according to geographic region, nodal status, centrally assessed hormonal receptor status and type of anthracycline.
Groups:
- Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane: Trastuzumab and pertuzumab were administered concurrently for up to a total duration of 1 year (up to 18 cycles [1 Cycle = 21 days]) with the taxane (docetaxel or paclitaxel) component of chemotherapy following anthracycline [5 fluorouracil, epirubicin, and cyclophosphamide (FEC) or epirubicin and cyclophosphamide (EC) or doxorubicin and cyclophosphamide (AC)] based chemotherapy.
- Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab: Trastuzumab emtansine and pertuzumab continued for up to a total duration of 1 year (up to 18 cycles [1 Cycle = 21 days]) following anthracycline [5 fluorouracil, epirubicin, and cyclophosphamide (FEC) or epirubicin and cyclophosphamide (EC) or doxorubicin and cyclophosphamide (AC)] based chemotherapy.
Period: Overall Study
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Started | 918 | 928
Completed | 0 | 0 (There is a difference in the death count displayed here and in the All-Cause Mortality section under Adverse Events. The difference relates to a participant that died and who was randomized to the AC-KP arm, but never received trastuzumab emtansine. Consequently they were assigned to the AC-THP for safety analyses. This death counts in the AC-KP arm when summary is based on the ITT population, but counts in the AC-THP arm when the summary on the safety population.)
Not Completed | 918 | 928
Not completed — Death | 44 | 56
Not completed — Lost to Follow-up | 46 | 39
Not completed — Various reasons | 4 | 4
Not completed — Physician Decision | 7 | 5
Not completed — Study Terminated By Sponsor | 758 | 773
Not completed — Withdrawal by Subject | 59 | 51

BASELINE CHARACTERISTICS:
Population: Baseline Measures are based on the Intent-to-Treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab | Total
Number analyzed (Participants) | 918 | 928 | 1846
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (10.8) | 51.9 (10.8) | 51.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 913 | 926 | 1839
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 68 | 138
  Not Hispanic or Latino | 798 | 790 | 1588
  Unknown or Not Reported | 50 | 70 | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 12 | 24
  Asian | 267 | 275 | 542
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 15 | 8 | 23
  White | 558 | 565 | 1123
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 63 | 65 | 128

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-Free Survival (IDFS) in the Node-Positive Subpopulation
Description: IDFS event was defined as the time from randomization until the date of first occurrence of one of the following: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer [bc] involving the same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive bc recurrence (an invasive bc in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); Contralateral or ipsilateral second primary invasive bc; Distant recurrence (evidence of bc in any anatomic site [other than the three sites mentioned above]) that has either been histologically confirmed or clinically/radiographically diagnosed as recurrent invasive bc; Death attributable to any cause, including bc, non-bc, or unknown cause. 3-year IDFS event-free rate per randomized treatment arms in the ITT population was estimated using the Kaplan-Meier method and estimated the probability of a participant being event-free after 3 years after randomization.
Time Frame: Last participant randomized to data cut-off date of 27 November 2019 (approximately 70 months). The 3 year IDFS event-free rate was assessed based on the data collected for each participant considering the cut-off date mentioned above.
Population: The ITT lymph node positive population was a subpopulation of the randomized participant population including patients with positive lymph node.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 826 | 832
Percent Probability | 94.10 [92.46 to 95.73] | 92.75 [90.95 to 94.54]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.8270, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI [0.71 to 1.32]

2. Primary Outcome: Invasive Disease-Free Survival (IDFS) in the Overall Population
Description: IDFS event was defined as the time from randomization until the date of first occurrence of one of the following: Ipsilateral invasive breast tumor recurrence (an invasive breast cancer [bc] involving the same breast parenchyma as the original primary lesion); Ipsilateral local-regional invasive bc recurrence (an invasive bc in the axilla, regional lymph nodes, chest wall, and/or skin of the ipsilateral breast); Contralateral or ipsilateral second primary invasive bc; Distant recurrence (evidence of bc in any anatomic site [other than the three sites mentioned above]) that has either been histologically confirmed or clinically/radiographically diagnosed as recurrent invasive bc; Death attributable to any cause, including bc, non-bc, or unknown cause. 3-year IDFS event-free rate per randomized treatment arms in the ITT population were estimated using the Kaplan-Meier method and estimated the probability of a patient being event-free after 3 years after randomization.
Time Frame: First participant randomized up to approximately 7.5 years
Population: The ITT Population comprised all randomized patients, whether or not they received any study treatment or completed a full course of study treatment. Patients were analyzed according to their randomized treatment.
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 918 | 928
Percent Probability | 94.22 [92.68 to 95.76] | 93.06 [91.40 to 94.73]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.9291, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI [0.77 to 1.34]

3. Secondary Outcome: IDFS Plus Second Primary Non-Breast Cancer
Description: IDFS including second primary non-breast cancer was defined the same way as IDFS for the primary endpoint but including second primary non breast invasive cancer as an event (with the exception of non-melanoma skin cancers and carcinoma in situ (CIS) of any site).
Time Frame: Baseline up to approximately 70 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 918 | 928
Percent Probability | 93.43 [91.79 to 95.06] | 92.26 [90.51 to 94.02]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.8756, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI [0.74 to 1.30]

4. Secondary Outcome: Disease-Free Survival (DFS)
Description: DFS was defined as time between randomization and first occurrence of IDFS, second primary non-breast cancer and contralateral or ipsilateral ductal carcinoma in situ (DCIS).
Time Frame: Baseline up to approximately 70 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 918 | 928
Percent Probability | 93.32 [91.67 to 94.97] | 92.04 [90.26 to 93.81]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.9341, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI [0.75 to 1.31]

5. Secondary Outcome: Distant Recurrence-Free Interval (DRFI)
Description: DRFI was defined as time between randomization and first occurrence of distant breast cancer recurrence.
Time Frame: Baseline up to approximately 70 months
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 918 | 928
Percent Probability | 95.23 [93.82 to 96.64] | 94.91 [93.46 to 96.36]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.4577, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI [0.61 to 1.25]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: First participant randomized up to approximately 7.5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 918 | 928
Percent Probability | 96.03 [94.72 to 97.34] | 94.86 [93.40 to 96.32]
Statistical Analysis 1: Comparison: Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane vs Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab; Test type: Superiority; p = 0.2864, Log Rank; Hazard Ratio (HR) = 1.24, 95% CI [0.83 to 1.84]

7. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. AEs were reported based on the national cancer institute common terminology criteria for AEs, Version 4.0 (NCI-CTCAE, v4.0).
Time Frame: From randomization to approximately 7.5 years
Population: The safety population included all randomized participants who received at least one full or partial dose of any study treatment. 8 participants were randomized but did not receive any study treatment (5 in the Anthracycline, Trastuzumab, Pertuzumab, and Taxane [AC-THP] arm, 3 in the Anthracycline, Trastuzumab Emtansine and Pertuzumab [AC-KP] arm). 16 participants in the AC-THP and 13 participants in the AC-KP arm only received AC but no HER2 targeted therapy and were assigned to the AC-THP arm.
Measure: Number; unit: Percentage of participants
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 926 | 912
Percentage of participants | 98.5 | 99.1

8. Secondary Outcome: Percentage of Participants With Decrease in Left Ventricular Ejection Fraction (LVEF) From Baseline Over Time
Description: LVEF was assessed using either echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans.
Time Frame: First participant randomized up to approximately 7.5 years.
Population: The safety population included all randomized participants who received at least one full or partial dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 926 | 912
Participants
  Decrease from baseline <10 Ejection Fraction (EF) points: number analyzed (Participants) | 914 | 912
  Decrease from baseline <10 Ejection Fraction (EF) points | 506 | 522
  Absolute value >= 50% and decrease from baseline >= 10 EF points: number analyzed (Participants) | 914 | 912
  Absolute value >= 50% and decrease from baseline >= 10 EF points | 254 | 245
  Absolute value < 50% and decrease from baseline >= 10 EF points: number analyzed (Participants) | 914 | 912
  Absolute value < 50% and decrease from baseline >= 10 EF points | 71 | 35
  Absolute value < 50% and decrease from baseline >= 15 EF points: number analyzed (Participants) | 914 | 912
  Absolute value < 50% and decrease from baseline >= 15 EF points | 61 | 28

9. Secondary Outcome: European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Score
Description: The EORTC QLQ-C30 included global health status, functional scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea/vomiting, and pain) and single items (dyspnoea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at all' to 4 'Very much'; 2 questions used 7-point scale [1 'very poor' to 7 'Excellent']). Scores were averaged and transformed to 0 - 100 scale, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms, with changes of 7 - 15 points considered to be a clinically meaningful detioration to participants. A positive value means an increase, while a negative value means a decrease, in score at the indicated time-point relative to the score at baseline (Cycle 1, Day 1).
Time Frame: Baseline, Cycles 1, 2, 3, 4, 5, 9, 14, End of Treatment, Follow-up Month 6, Follow-up Month 12, Follow-up Month 18
Population: The Patient Reported Outcome (PRO) Population includes participants with both a baseline assessment and at least one post-baseline assessment in any PRO items. The variation of the number of participants in the table reflects the number of participants with corresponding scores at the given visits and at baseline.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 869 | 891
Units on a Scale
  Baseline: Appetite Loss: number analyzed (Participants) | 869 | 888
  Baseline: Appetite Loss | 8.2 (17.6) | 7.6 (16.8)
  Change at Cycle 1: Appetite Loss: number analyzed (Participants) | 835 | 857
  Change at Cycle 1: Appetite Loss | 12.2 (27.9) | 10.8 (26.6)
  Change at Cycle 2: Appetite Loss: number analyzed (Participants) | 816 | 827
  Change at Cycle 2: Appetite Loss | 15.2 (27.7) | 13.1 (26.7)
  Change at Cycle 3: Appetite Loss: number analyzed (Participants) | 816 | 833
  Change at Cycle 3: Appetite Loss | 14.3 (28.2) | 10.3 (25.7)
  Change at Cycle 4: Appetite Loss: number analyzed (Participants) | 815 | 834
  Change at Cycle 4: Appetite Loss | 16.2 (29.8) | 9.4 (25.5)
  Change at Cycle 5: Appetite Loss: number analyzed (Participants) | 814 | 826
  Change at Cycle 5: Appetite Loss | 12.0 (28.4) | 9.0 (26.2)
  Change at Cycle 9: Appetite Loss: number analyzed (Participants) | 792 | 792
  Change at Cycle 9: Appetite Loss | 5.7 (23.9) | 8.2 (25.7)
  Change at Cycle 14: Appetite Loss: number analyzed (Participants) | 772 | 750
  Change at Cycle 14: Appetite Loss | 2.2 (23.1) | 6.4 (25.4)
  Change at EoT: Appetite Loss: number analyzed (Participants) | 806 | 810
  Change at EoT: Appetite Loss | 0.5 (22.3) | 5.6 (25.1)
  Change at FU Month 6: Appetite Loss: number analyzed (Participants) | 766 | 744
  Change at FU Month 6: Appetite Loss | -1.3 (20.7) | -2.4 (20.3)
  Change at FU Month 12: Appetite Loss: number analyzed (Participants) | 738 | 722
  Change at FU Month 12: Appetite Loss | -2.2 (20.8) | -2.3 (20.5)
  Change at FU Month 18: Appetite Loss: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Appetite Loss |  | -16.7 (23.6)
  Baseline: Constipation: number analyzed (Participants) | 869 | 884
  Baseline: Constipation | 9.6 (19.4) | 9.0 (19.6)
  Change at Cycle 1: Constipation: number analyzed (Participants) | 835 | 855
  Change at Cycle 1: Constipation | 8.4 (22.5) | 8.0 (26.1)
  Change at Cycle 2: Constipation: number analyzed (Participants) | 812 | 821
  Change at Cycle 2: Constipation | 1.1 (25.0) | 0.9 (23.1)
  Change at Cycle 3: Constipation: number analyzed (Participants) | 812 | 829
  Change at Cycle 3: Constipation | 2.0 (24.6) | 0.2 (22.2)
  Change at Cycle 4: Constipation: number analyzed (Participants) | 811 | 829
  Change at Cycle 4: Constipation | 2.5 (24.3) | -0.6 (23.2)
  Change at Cycle 5: Constipation: number analyzed (Participants) | 813 | 820
  Change at Cycle 5: Constipation | 0.5 (22.4) | -0.4 (22.1)
  Change at Cycle 9: Constipation: number analyzed (Participants) | 792 | 788
  Change at Cycle 9: Constipation | -0.7 (21.7) | 3.3 (24.7)
  Change at Cycle 14: Constipation: number analyzed (Participants) | 772 | 743
  Change at Cycle 14: Constipation | 0.6 (21.1) | 4.2 (24.6)
  Change at EoT: Constipation: number analyzed (Participants) | 805 | 805
  Change at EoT: Constipation | 0.2 (21.8) | 4.7 (25.1)
  Change at FU Month 6: Constipation: number analyzed (Participants) | 766 | 742
  Change at FU Month 6: Constipation | 3.4 (23.2) | 1.5 (24.1)
  Change at FU Month 12: Constipation: number analyzed (Participants) | 740 | 719
  Change at FU Month 12: Constipation | 2.8 (22.8) | 2.0 (23.3)
  Change at FU Month 18: Constipation: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Constipation |  | 0.0 (0.0)
  Baseline: Diarrhea: number analyzed (Participants) | 864 | 878
  Baseline: Diarrhea | 5.2 (13.2) | 4.7 (12.9)
  Change at Cycle 1: Diarrhea: number analyzed (Participants) | 832 | 848
  Change at Cycle 1: Diarrhea | 4.7 (20.3) | 4.2 (18.4)
  Change at Cycle 2: Diarrhea: number analyzed (Participants) | 813 | 815
  Change at Cycle 2: Diarrhea | 32.5 (32.8) | 16.0 (26.9)
  Change at Cycle 3: Diarrhea: number analyzed (Participants) | 814 | 824
  Change at Cycle 3: Diarrhea | 28.4 (30.5) | 11.3 (23.5)
  Change at Cycle 4: Diarrhea: number analyzed (Participants) | 810 | 824
  Change at Cycle 4: Diarrhea | 26.5 (30.0) | 10.3 (23.6)
  Change at Cycle 5: Diarrhea: number analyzed (Participants) | 808 | 815
  Change at Cycle 5: Diarrhea | 23.9 (30.4) | 8.8 (22.8)
  Change at Cycle 9: Diarrhea: number analyzed (Participants) | 788 | 786
  Change at Cycle 9: Diarrhea | 12.6 (24.6) | 4.7 (21.7)
  Change at Cycle 14: Diarrhea: number analyzed (Participants) | 767 | 740
  Change at Cycle 14: Diarrhea | 12.5 (26.4) | 5.1 (20.3)
  Change at EoT: Diarrhea: number analyzed (Participants) | 805 | 798
  Change at EoT: Diarrhea | 10.3 (25.2) | 3.0 (19.4)
  Change at FU Month 6: Diarrhea: number analyzed (Participants) | 759 | 734
  Change at FU Month 6: Diarrhea | -0.3 (16.4) | -1.1 (16.3)
  Change at FU Month 12: Diarrhea: number analyzed (Participants) | 732 | 712
  Change at FU Month 12: Diarrhea | -0.3 (17.8) | 0.0 (17.1)
  Change at FU Month 18: Diarrhea: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Diarrhea |  | -16.7 (23.6)
  Baseline: Dyspnea: number analyzed (Participants) | 869 | 887
  Baseline: Dyspnea | 5.8 (14.0) | 6.2 (14.3)
  Change at Cycle 1: Dyspnea: number analyzed (Participants) | 838 | 856
  Change at Cycle 1: Dyspnea | 10.4 (21.4) | 9.2 (21.8)
  Change at Cycle 2: Dyspnea: number analyzed (Participants) | 816 | 825
  Change at Cycle 2: Dyspnea | 11.6 (22.0) | 7.4 (20.6)
  Change at Cycle 3: Dyspnea: number analyzed (Participants) | 817 | 833
  Change at Cycle 3: Dyspnea | 13.4 (23.2) | 6.5 (20.5)
  Change at Cycle 4: Dyspnea: number analyzed (Participants) | 816 | 833
  Change at Cycle 4: Dyspnea | 14.3 (23.7) | 5.9 (20.8)
  Change at Cycle 5: Dyspnea: number analyzed (Participants) | 816 | 826
  Change at Cycle 5: Dyspnea | 13.7 (22.4) | 5.6 (19.8)
  Change at Cycle 9: Dyspnea: number analyzed (Participants) | 790 | 792
  Change at Cycle 9: Dyspnea | 7.8 (19.3) | 7.5 (21.4)
  Change at Cycle 14: Dyspnea: number analyzed (Participants) | 773 | 750
  Change at Cycle 14: Dyspnea | 6.8 (20.8) | 8.1 (21.6)
  Change at EoT: Dyspnea: number analyzed (Participants) | 805 | 809
  Change at EoT: Dyspnea | 7.6 (21.1) | 8.8 (22.3)
  Change at FU Month 6: Dyspnea: number analyzed (Participants) | 766 | 743
  Change at FU Month 6: Dyspnea | 7.0 (20.8) | 5.3 (19.7)
  Change at FU Month 12: Dyspnea: number analyzed (Participants) | 740 | 722
  Change at FU Month 12: Dyspnea | 6.2 (20.9) | 5.8 (20.5)
  Change at FU Month 18: Dyspnea: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Dyspnea |  | -16.7 (23.6)
  Baseline: Fatigue: number analyzed (Participants) | 868 | 887
  Baseline: Fatigue | 21.5 (18.6) | 20.6 (18.6)
  Change at Cycle 1: Fatigue: number analyzed (Participants) | 837 | 857
  Change at Cycle 1: Fatigue | 13.2 (21.5) | 14.4 (22.1)
  Change at Cycle 2: Fatigue: number analyzed (Participants) | 815 | 825
  Change at Cycle 2: Fatigue | 15.4 (22.7) | 11.2 (21.7)
  Change at Cycle 3: Fatigue: number analyzed (Participants) | 816 | 833
  Change at Cycle 3: Fatigue | 15.3 (23.1) | 8.7 (20.9)
  Change at Cycle 4: Fatigue: number analyzed (Participants) | 816 | 834
  Change at Cycle 4: Fatigue | 16.0 (23.4) | 8.2 (20.7)
  Change at Cycle 5: Fatigue: number analyzed (Participants) | 815 | 826
  Change at Cycle 5: Fatigue | 14.9 (22.8) | 8.4 (21.1)
  Change at Cycle 9: Fatigue: number analyzed (Participants) | 790 | 791
  Change at Cycle 9: Fatigue | 8.4 (22.0) | 9.8 (20.8)
  Change at Cycle 14: Fatigue: number analyzed (Participants) | 772 | 751
  Change at Cycle 14: Fatigue | 6.7 (22.0) | 10.6 (22.4)
  Change at EoT: Fatigue: number analyzed (Participants) | 808 | 809
  Change at EoT: Fatigue | 5.5 (22.9) | 9.3 (21.9)
  Change at FU Month 6: Fatigue: number analyzed (Participants) | 765 | 744
  Change at FU Month 6: Fatigue | 2.8 (21.9) | 3.1 (21.9)
  Change at FU Month 12: Fatigue: number analyzed (Participants) | 739 | 722
  Change at FU Month 12: Fatigue | 1.9 (22.1) | 1.8 (20.8)
  Change at FU Month 18: Fatigue: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Fatigue |  | -5.6 (39.3)
  Baseline: Financial Difficulties: number analyzed (Participants) | 859 | 876
  Baseline: Financial Difficulties | 20.1 (28.3) | 19.9 (28.5)
  Change at Cycle 1: Financial Difficulties: number analyzed (Participants) | 825 | 843
  Change at Cycle 1: Financial Difficulties | 2.2 (25.2) | 0.3 (24.8)
  Change at Cycle 2: Financial Difficulties: number analyzed (Participants) | 808 | 810
  Change at Cycle 2: Financial Difficulties | 2.0 (25.7) | -0.6 (25.3)
  Change at Cycle 3: Financial Difficulties: number analyzed (Participants) | 810 | 820
  Change at Cycle 3: Financial Difficulties | 3.9 (24.7) | -0.4 (25.0)
  Change at Cycle 4: Financial Difficulties: number analyzed (Participants) | 802 | 820
  Change at Cycle 4: Financial Difficulties | 3.7 (24.9) | -0.2 (25.4)
  Change at Cycle 5: Financial Difficulties: number analyzed (Participants) | 801 | 811
  Change at Cycle 5: Financial Difficulties | 3.4 (25.3) | 0.7 (26.2)
  Change at Cycle 9: Financial Difficulties: number analyzed (Participants) | 784 | 782
  Change at Cycle 9: Financial Difficulties | 0.9 (25.6) | -0.5 (26.6)
  Change at Cycle 14: Financial Difficulties: number analyzed (Participants) | 763 | 736
  Change at Cycle 14: Financial Difficulties | -1.4 (25.1) | -1.0 (27.2)
  Change at EoT: Financial Difficulties: number analyzed (Participants) | 799 | 797
  Change at EoT: Financial Difficulties | -1.1 (27.3) | -1.7 (25.7)
  Change at FU Month 6: Financial Difficulties: number analyzed (Participants) | 755 | 732
  Change at FU Month 6: Financial Difficulties | -3.8 (27.4) | -5.2 (28.7)
  Change at FU Month 12: Financial Difficulties: number analyzed (Participants) | 728 | 708
  Change at FU Month 12: Financial Difficulties | -5.1 (28.6) | -6.8 (28.3)
  Change at FU Month 18: Financial Difficulties: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Financial Difficulties |  | 0.0 (0.0)
  Baseline: Insomnia: number analyzed (Participants) | 869 | 888
  Baseline: Insomnia | 23.9 (26.1) | 24.9 (27.6)
  Change at Cycle 1: Insomnia: number analyzed (Participants) | 838 | 857
  Change at Cycle 1: Insomnia | 3.6 (30.2) | 1.8 (28.8)
  Change at Cycle 2: Insomnia: number analyzed (Participants) | 816 | 828
  Change at Cycle 2: Insomnia | 6.0 (30.5) | 0.4 (30.0)
  Change at Cycle 3: Insomnia: number analyzed (Participants) | 815 | 835
  Change at Cycle 3: Insomnia | 6.2 (30.2) | -0.1 (30.3)
  Change at Cycle 4: Insomnia: number analyzed (Participants) | 817 | 835
  Change at Cycle 4: Insomnia | 8.6 (31.3) | 1.1 (30.4)
  Change at Cycle 5: Insomnia: number analyzed (Participants) | 814 | 827
  Change at Cycle 5: Insomnia | 5.2 (31.1) | 1.1 (29.9)
  Change at Cycle 9: Insomnia: number analyzed (Participants) | 790 | 791
  Change at Cycle 9: Insomnia | 4.3 (30.5) | 1.1 (29.9)
  Change at Cycle 14: Insomnia: number analyzed (Participants) | 773 | 751
  Change at Cycle 14: Insomnia | 2.7 (30.6) | 2.7 (30.2)
  Change at EoT: Insomnia: number analyzed (Participants) | 807 | 810
  Change at EoT: Insomnia | 2.5 (30.8) | 0.9 (30.2)
  Change at FU Month 6: Insomnia: number analyzed (Participants) | 765 | 744
  Change at FU Month 6: Insomnia | 0.9 (29.5) | -2.3 (29.6)
  Change at FU Month 12: Insomnia: number analyzed (Participants) | 739 | 724
  Change at FU Month 12: Insomnia | 0.0 (30.2) | -2.9 (30.4)
  Change at FU Month 18: Insomnia: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Insomnia |  | -16.7 (23.6)
  Baseline: Nausea/Vomiting: number analyzed (Participants) | 869 | 887
  Baseline: Nausea/Vomiting | 2.6 (9.4) | 2.3 (7.1)
  Change at Cycle 1: Nausea/Vomiting: number analyzed (Participants) | 839 | 856
  Change at Cycle 1: Nausea/Vomiting | 10.4 (19.5) | 10.5 (17.8)
  Change at Cycle 2: Nausea/Vomiting: number analyzed (Participants) | 816 | 827
  Change at Cycle 2: Nausea/Vomiting | 6.0 (16.5) | 7.5 (16.1)
  Change at Cycle 3: Nausea/Vomiting: number analyzed (Participants) | 817 | 833
  Change at Cycle 3: Nausea/Vomiting | 5.0 (16.2) | 5.2 (13.9)
  Change at Cycle 4: Nausea/Vomiting: number analyzed (Participants) | 816 | 834
  Change at Cycle 4: Nausea/Vomiting | 4.7 (16.0) | 3.7 (12.8)
  Change at Cycle 5: Nausea/Vomiting: number analyzed (Participants) | 817 | 826
  Change at Cycle 5: Nausea/Vomiting | 4.0 (15.6) | 3.2 (13.1)
  Change at Cycle 9: Nausea/Vomiting: number analyzed (Participants) | 792 | 792
  Change at Cycle 9: Nausea/Vomiting | 1.1 (13.8) | 2.8 (11.5)
  Change at Cycle 14: Nausea/Vomiting: number analyzed (Participants) | 773 | 751
  Change at Cycle 14: Nausea/Vomiting | 1.1 (12.3) | 3.0 (12.1)
  Change at EoT: Nausea/Vomiting: number analyzed (Participants) | 806 | 809
  Change at EoT: Nausea/Vomiting | 0.9 (13.2) | 1.7 (12.0)
  Change at FU Month 6: Nausea/Vomiting: number analyzed (Participants) | 766 | 744
  Change at FU Month 6: Nausea/Vomiting | 0.2 (11.6) | 0.1 (10.1)
  Change at FU Month 12: Nausea/Vomiting: number analyzed (Participants) | 740 | 721
  Change at FU Month 12: Nausea/Vomiting | 0.5 (12.4) | 0.6 (10.3)
  Change at FU Month 18: Nausea/Vomiting: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Nausea/Vomiting |  | -8.3 (11.8)
  Baseline: Pain: number analyzed (Participants) | 869 | 889
  Baseline: Pain | 17.4 (20.1) | 16.4 (20.0)
  Change at Cycle 1: Pain: number analyzed (Participants) | 839 | 859
  Change at Cycle 1: Pain | 1.8 (22.8) | 1.1 (22.5)
  Change at Cycle 2: Pain: number analyzed (Participants) | 816 | 828
  Change at Cycle 2: Pain | 5.0 (24.5) | 2.8 (23.1)
  Change at Cycle 3: Pain: number analyzed (Participants) | 818 | 836
  Change at Cycle 3: Pain | 3.5 (23.7) | 2.5 (22.6)
  Change at Cycle 4: Pain: number analyzed (Participants) | 817 | 836
  Change at Cycle 4: Pain | 5.4 (23.2) | 3.1 (23.5)
  Change at Cycle 5: Pain: number analyzed (Participants) | 817 | 828
  Change at Cycle 5: Pain | 5.2 (23.7) | 3.8 (23.5)
  Change at Cycle 9: Pain: number analyzed (Participants) | 791 | 792
  Change at Cycle 9: Pain | 3.4 (22.6) | 3.9 (23.3)
  Change at Cycle 14: Pain: number analyzed (Participants) | 773 | 753
  Change at Cycle 14: Pain | 2.0 (23.4) | 5.7 (24.1)
  Change at EoT: Pain: number analyzed (Participants) | 809 | 812
  Change at EoT: Pain | 1.9 (23.3) | 5.1 (24.5)
  Change at FU Month 6: Pain: number analyzed (Participants) | 766 | 746
  Change at FU Month 6: Pain | 0.8 (23.0) | 1.4 (22.6)
  Change at FU Month 12: Pain: number analyzed (Participants) | 741 | 725
  Change at FU Month 12: Pain | 0.0 (23.3) | 0.5 (21.5)
  Change at FU Month 18: Pain: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Pain |  | -25.0 (35.4)
  Baseline: Cognitive Functioning: number analyzed (Participants) | 864 | 879
  Baseline: Cognitive Functioning | 88.6 (16.9) | 88.7 (16.3)
  Change at Cycle 1: Cognitive Functioning: number analyzed (Participants) | 832 | 851
  Change at Cycle 1: Cognitive Functioning | -9.7 (20.8) | -6.9 (19.3)
  Change at Cycle 2: Cognitive Functioning: number analyzed (Participants) | 813 | 818
  Change at Cycle 2: Cognitive Functioning | -9.4 (20.0) | -6.8 (19.3)
  Change at Cycle 3: Cognitive Functioning: number analyzed (Participants) | 814 | 824
  Change at Cycle 3: Cognitive Functioning | -10.1 (20.8) | -6.4 (19.4)
  Change at Cycle 4: Cognitive Functioning: number analyzed (Participants) | 810 | 825
  Change at Cycle 4: Cognitive Functioning | -11.8 (21.6) | -6.9 (19.6)
  Change at Cycle 5: Cognitive Functioning: number analyzed (Participants) | 807 | 816
  Change at Cycle 5: Cognitive Functioning | -10.8 (21.6) | -7.3 (20.3)
  Change at Cycle 9: Cognitive Functioning: number analyzed (Participants) | 789 | 787
  Change at Cycle 9: Cognitive Functioning | -8.3 (20.2) | -7.6 (20.1)
  Change at Cycle 14: Cognitive Functioning: number analyzed (Participants) | 768 | 742
  Change at Cycle 14: Cognitive Functioning | -8.1 (20.3) | -8.1 (20.6)
  Change at EoT: Cognitive Functioning: number analyzed (Participants) | 805 | 800
  Change at EoT: Cognitive Functioning | -8.7 (22.3) | -8.4 (20.9)
  Change at FU Month 6: Cognitive Functioning: number analyzed (Participants) | 760 | 735
  Change at FU Month 6: Cognitive Functioning | -8.0 (20.4) | -6.1 (19.7)
  Change at FU Month 12: Cognitive Functioning: number analyzed (Participants) | 733 | 713
  Change at FU Month 12: Cognitive Functioning | -7.1 (22.5) | -6.0 (20.7)
  Change at FU Month 18: Cognitive Functioning: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Cognitive Functioning |  | 16.7 (23.6)
  Baseline: Emotional Functioning: number analyzed (Participants) | 864 | 880
  Baseline: Emotional Functioning | 76.0 (19.7) | 75.7 (20.9)
  Change at Cycle 1: Emotional Functioning: number analyzed (Participants) | 832 | 849
  Change at Cycle 1: Emotional Functioning | -1.1 (20.3) | 0.0 (19.2)
  Change at Cycle 2: Emotional Functioning: number analyzed (Participants) | 813 | 819
  Change at Cycle 2: Emotional Functioning | -1.0 (20.8) | 1.6 (19.7)
  Change at Cycle 3: Emotional Functioning: number analyzed (Participants) | 814 | 825
  Change at Cycle 3: Emotional Functioning | -0.9 (21.2) | 2.2 (19.6)
  Change at Cycle 4: Emotional Functioning: number analyzed (Participants) | 810 | 826
  Change at Cycle 4: Emotional Functioning | -2.5 (22.3) | 2.8 (20.0)
  Change at Cycle 5: Emotional Functioning: number analyzed (Participants) | 808 | 817
  Change at Cycle 5: Emotional Functioning | -1.2 (22.2) | 2.6 (21.1)
  Change at Cycle 9: Emotional Functioning: number analyzed (Participants) | 789 | 788
  Change at Cycle 9: Emotional Functioning | 3.1 (20.9) | 2.9 (21.1)
  Change at Cycle 14: Emotional Functioning: number analyzed (Participants) | 768 | 743
  Change at Cycle 14: Emotional Functioning | 4.1 (21.0) | 2.5 (21.3)
  Change at EoT: Emotional Functioning: number analyzed (Participants) | 806 | 801
  Change at EoT: Emotional Functioning | 3.0 (22.4) | 3.1 (21.3)
  Change at FU Month 6: Emotional Functioning: number analyzed (Participants) | 760 | 736
  Change at FU Month 6: Emotional Functioning | 4.7 (21.2) | 6.1 (21.8)
  Change at FU Month 12: Emotional Functioning: number analyzed (Participants) | 733 | 714
  Change at FU Month 12: Emotional Functioning | 5.8 (22.1) | 6.5 (21.9)
  Change at FU Month 18: Emotional Functioning: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Emotional Functioning |  | 12.5 (17.7)
  Baseline: Physical Functioning: number analyzed (Participants) | 869 | 889
  Baseline: Physical Functioning | 88.4 (13.5) | 89.1 (12.3)
  Change at Cycle 1: Physical Functioning: number analyzed (Participants) | 838 | 859
  Change at Cycle 1: Physical Functioning | -6.0 (14.5) | -5.9 (13.4)
  Change at Cycle 2: Physical Functioning: number analyzed (Participants) | 816 | 827
  Change at Cycle 2: Physical Functioning | -7.8 (15.8) | -4.8 (12.8)
  Change at Cycle 3: Physical Functioning: number analyzed (Participants) | 817 | 835
  Change at Cycle 3: Physical Functioning | -7.1 (15.4) | -4.1 (13.0)
  Change at Cycle 4: Physical Functioning: number analyzed (Participants) | 816 | 835
  Change at Cycle 4: Physical Functioning | -8.4 (16.2) | -3.5 (13.1)
  Change at Cycle 5: Physical Functioning: number analyzed (Participants) | 817 | 827
  Change at Cycle 5: Physical Functioning | -8.3 (16.1) | -3.5 (13.3)
  Change at Cycle 9: Physical Functioning: number analyzed (Participants) | 789 | 793
  Change at Cycle 9: Physical Functioning | -4.0 (15.0) | -3.8 (14.2)
  Change at Cycle 14: Physical Functioning: number analyzed (Participants) | 773 | 752
  Change at Cycle 14: Physical Functioning | -2.7 (14.2) | -4.2 (14.2)
  Change at EoT: Physical Functioning: number analyzed (Participants) | 805 | 810
  Change at EoT: Physical Functioning | -2.2 (14.7) | -4.9 (15.0)
  Change at FU Month 6: Physical Functioning: number analyzed (Participants) | 766 | 747
  Change at FU Month 6: Physical Functioning | -0.6 (14.4) | -1.6 (13.6)
  Change at FU Month 12: Physical Functioning: number analyzed (Participants) | 739 | 724
  Change at FU Month 12: Physical Functioning | -0.1 (15.4) | -0.8 (13.2)
  Change at FU Month 18: Physical Functioning: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Physical Functioning |  | 13.3 (18.9)
  Baseline: Role Functioning: number analyzed (Participants) | 869 | 889
  Baseline: Role Functioning | 83.1 (21.7) | 83.4 (21.3)
  Change at Cycle 1: Role Functioning: number analyzed (Participants) | 837 | 859
  Change at Cycle 1: Role Functioning | -5.1 (24.5) | -5.7 (24.9)
  Change at Cycle 2: Role Functioning: number analyzed (Participants) | 816 | 828
  Change at Cycle 2: Role Functioning | -9.7 (26.6) | -5.5 (24.0)
  Change at Cycle 3: Role Functioning: number analyzed (Participants) | 817 | 835
  Change at Cycle 3: Role Functioning | -8.9 (26.7) | -2.7 (23.2)
  Change at Cycle 4: Role Functioning: number analyzed (Participants) | 815 | 836
  Change at Cycle 4: Role Functioning | -10.7 (27.5) | -3.2 (23.7)
  Change at Cycle 5: Role Functioning: number analyzed (Participants) | 817 | 827
  Change at Cycle 5: Role Functioning | -9.4 (27.3) | -3.5 (23.9)
  Change at Cycle 9: Role Functioning: number analyzed (Participants) | 792 | 792
  Change at Cycle 9: Role Functioning | -3.3 (25.4) | -3.2 (24.1)
  Change at Cycle 14: Role Functioning: number analyzed (Participants) | 772 | 752
  Change at Cycle 14: Role Functioning | -0.5 (25.0) | -4.3 (25.3)
  Change at EoT: Role Functioning: number analyzed (Participants) | 806 | 811
  Change at EoT: Role Functioning | -0.2 (26.3) | -3.5 (24.9)
  Change at FU Month 6: Role Functioning: number analyzed (Participants) | 766 | 746
  Change at FU Month 6: Role Functioning | 2.2 (24.7) | 2.4 (24.1)
  Change at FU Month 12: Role Functioning: number analyzed (Participants) | 740 | 724
  Change at FU Month 12: Role Functioning | 2.6 (25.9) | 3.7 (23.8)
  Change at FU Month 18: Role Functioning: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Role Functioning |  | 8.3 (11.8)
  Baseline: Social Functioning: number analyzed (Participants) | 863 | 877
  Baseline: Social Functioning | 83.0 (22.9) | 83.2 (21.6)
  Change at Cycle 1: Social Functioning: number analyzed (Participants) | 831 | 849
  Change at Cycle 1: Social Functioning | -8.0 (24.3) | -5.3 (22.8)
  Change at Cycle 2: Social Functioning: number analyzed (Participants) | 812 | 816
  Change at Cycle 2: Social Functioning | -10.1 (26.1) | -4.1 (23.6)
  Change at Cycle 3: Social Functioning: number analyzed (Participants) | 814 | 823
  Change at Cycle 3: Social Functioning | -9.5 (25.6) | -3.3 (24.4)
  Change at Cycle 4: Social Functioning: number analyzed (Participants) | 808 | 823
  Change at Cycle 4: Social Functioning | -10.3 (26.3) | -3.2 (24.2)
  Change at Cycle 5: Social Functioning: number analyzed (Participants) | 808 | 815
  Change at Cycle 5: Social Functioning | -8.7 (26.5) | -2.6 (23.7)
  Change at Cycle 9: Social Functioning: number analyzed (Participants) | 789 | 785
  Change at Cycle 9: Social Functioning | -1.7 (25.1) | -3.4 (24.9)
  Change at Cycle 14: Social Functioning: number analyzed (Participants) | 768 | 738
  Change at Cycle 14: Social Functioning | -0.1 (25.3) | -2.4 (24.9)
  Change at EoT: Social Functioning: number analyzed (Participants) | 804 | 798
  Change at EoT: Social Functioning | 0.3 (26.1) | -1.6 (24.1)
  Change at FU Month 6: Social Functioning: number analyzed (Participants) | 759 | 733
  Change at FU Month 6: Social Functioning | 3.3 (24.8) | 4.0 (24.7)
  Change at FU Month 12: Social Functioning: number analyzed (Participants) | 732 | 711
  Change at FU Month 12: Social Functioning | 4.6 (25.2) | 6.4 (22.7)
  Change at FU Month 18: Social Functioning: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Social Functioning |  | 33.3 (47.1)
  Baseline: Global Health Status: number analyzed (Participants) | 863 | 878
  Baseline: Global Health Status | 74.3 (18.7) | 73.9 (18.7)
  Change at Cycle 1: Global Health Status: number analyzed (Participants) | 831 | 850
  Change at Cycle 1: Global Health Status | -7.5 (20.1) | -7.2 (20.4)
  Change at Cycle 2: Global Health Status: number analyzed (Participants) | 812 | 815
  Change at Cycle 2: Global Health Status | -12.4 (22.6) | -7.1 (20.2)
  Change at Cycle 3: Global Health Status: number analyzed (Participants) | 814 | 823
  Change at Cycle 3: Global Health Status | -11.7 (20.6) | -5.2 (19.1)
  Change at Cycle 4: Global Health Status: number analyzed (Participants) | 807 | 824
  Change at Cycle 4: Global Health Status | -12.7 (21.3) | -5.5 (19.6)
  Change at Cycle 5: Global Health Status: number analyzed (Participants) | 807 | 815
  Change at Cycle 5: Global Health Status | -12.1 (21.7) | -5.8 (19.7)
  Change at Cycle 9: Global Health Status: number analyzed (Participants) | 784 | 787
  Change at Cycle 9: Global Health Status | -5.9 (20.1) | -6.4 (20.6)
  Change at Cycle 14: Global Health Status: number analyzed (Participants) | 766 | 741
  Change at Cycle 14: Global Health Status | -3.9 (21.1) | -6.3 (20.8)
  Change at EoT: Global Health Status: number analyzed (Participants) | 804 | 798
  Change at EoT: Global Health Status | -3.5 (21.3) | -4.9 (20.7)
  Change at FU Month 6: Global Health Status: number analyzed (Participants) | 758 | 733
  Change at FU Month 6: Global Health Status | -0.6 (21.3) | 0.3 (21.4)
  Change at FU Month 12: Global Health Status: number analyzed (Participants) | 731 | 712
  Change at FU Month 12: Global Health Status | -0.2 (21.9) | 1.2 (20.8)
  Change at FU Month 18: Global Health Status: number analyzed (Participants) | 0 | 2
  Change at FU Month 18: Global Health Status |  | 16.7 (23.6)

10. Secondary Outcome: EORTC Quality of Life Questionnaire-Breast Cancer 23 (QLQ-BR23) Score
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30. There are four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Scores averaged and transformed to 0-100 scale. High score for functional scale indicated high/better level of functioning/healthy functioning. Higher scores for symptom scales represent higher levels of symptoms/problems. For functional scales, positive change from baseline indicated improvement in quality of life (QOL) while negative change from baseline indicated a deterioration. For symptom scales, positive change from baseline indicated deterioration and negative change indicated improvement.
Time Frame: Baseline, Cycles 1, 2, 3, 4, 5, 9, 14, End of Treatment, Follow-up Month 6, Follow-up Month 12, Follow-up Month 18
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 869 | 891
Units on a Scale
  Baseline: Arm Symptoms: number analyzed (Participants) | 844 | 861
  Baseline: Arm Symptoms | 19.9 (18.7) | 19.5 (18.4)
  Change at Cycle 1: Arm Symptoms: number analyzed (Participants) | 804 | 831
  Change at Cycle 1: Arm Symptoms | -1.3 (19.2) | -3.1 (18.7)
  Change at Cycle 2: Arm Symptoms: number analyzed (Participants) | 788 | 798
  Change at Cycle 2: Arm Symptoms | -2.8 (18.8) | -3.0 (18.7)
  Change at Cycle 3: Arm Symptoms: number analyzed (Participants) | 788 | 805
  Change at Cycle 3: Arm Symptoms | -3.5 (18.7) | -3.5 (18.1)
  Change at Cycle 4: Arm Symptoms: number analyzed (Participants) | 786 | 803
  Change at Cycle 4: Arm Symptoms | -2.0 (19.8) | -2.9 (19.2)
  Change at Cycle 5: Arm Symptoms: number analyzed (Participants) | 790 | 798
  Change at Cycle 5: Arm Symptoms | -0.5 (20.8) | -2.6 (19.8)
  Change at Cycle 9: Arm Symptoms: number analyzed (Participants) | 768 | 765
  Change at Cycle 9: Arm Symptoms | -0.2 (20.4) | -1.1 (19.6)
  Change at Cycle 14: Arm Symptoms: number analyzed (Participants) | 754 | 725
  Change at Cycle 14: Arm Symptoms | 0.3 (21.3) | 1.3 (21.8)
  Change at EoT: Arm Symptoms: number analyzed (Participants) | 784 | 785
  Change at EoT: Arm Symptoms | 0.1 (21.6) | 0.4 (21.7)
  Change at FU Month 6: Arm Symptoms: number analyzed (Participants) | 739 | 716
  Change at FU Month 6: Arm Symptoms | -0.1 (22.1) | -1.3 (20.0)
  Change at FU Month 12: Arm Symptoms: number analyzed (Participants) | 714 | 693
  Change at FU Month 12: Arm Symptoms | -0.8 (22.4) | -2.8 (20.5)
  Change at FU Month 18: Arm Symptoms: number analyzed (Participants) | 0 | 0
  Baseline: Breast Symptoms: number analyzed (Participants) | 843 | 859
  Baseline: Breast Symptoms | 17.5 (17.4) | 16.8 (16.3)
  Change at Cycle 1: Breast Symptoms: number analyzed (Participants) | 802 | 828
  Change at Cycle 1: Breast Symptoms | -2.3 (16.3) | -2.5 (16.2)
  Change at Cycle 2: Breast Symptoms: number analyzed (Participants) | 786 | 795
  Change at Cycle 2: Breast Symptoms | -3.3 (17.1) | -2.9 (16.7)
  Change at Cycle 3: Breast Symptoms: number analyzed (Participants) | 785 | 803
  Change at Cycle 3: Breast Symptoms | -4.0 (17.5) | -3.1 (16.5)
  Change at Cycle 4: Breast Symptoms: number analyzed (Participants) | 786 | 800
  Change at Cycle 4: Breast Symptoms | -3.9 (17.7) | -3.3 (17.4)
  Change at Cycle 5: Breast Symptoms: number analyzed (Participants) | 787 | 796
  Change at Cycle 5: Breast Symptoms | -3.1 (18.6) | -2.6 (18.2)
  Change at Cycle 9: Breast Symptoms: number analyzed (Participants) | 768 | 763
  Change at Cycle 9: Breast Symptoms | 1.7 (19.7) | 0.3 (17.5)
  Change at Cycle 14: Breast Symptoms: number analyzed (Participants) | 751 | 724
  Change at Cycle 14: Breast Symptoms | -0.2 (18.8) | 0.5 (19.1)
  Change at EoT: Breast Symptoms: number analyzed (Participants) | 781 | 783
  Change at EoT: Breast Symptoms | -1.0 (19.3) | 0.3 (18.8)
  Change at FU Month 6: Breast Symptoms: number analyzed (Participants) | 738 | 714
  Change at FU Month 6: Breast Symptoms | -2.5 (19.1) | -1.5 (18.4)
  Change at FU Month 12: Breast Symptoms: number analyzed (Participants) | 713 | 691
  Change at FU Month 12: Breast Symptoms | -4.2 (18.9) | -3.7 (18.0)
  Change at FU Month 18: Breast Symptoms: number analyzed (Participants) | 0 | 0
  Baseline: Systemic Therapy Side Effects (SE): number analyzed (Participants) | 845 | 868
  Baseline: Systemic Therapy Side Effects (SE) | 8.5 (9.9) | 8.7 (9.9)
  Change at Cycle 1: Systemic Therapy SE: number analyzed (Participants) | 812 | 838
  Change at Cycle 1: Systemic Therapy SE | 24.9 (17.3) | 23.3 (17.6)
  Change at Cycle 2: Systemic Therapy SE: number analyzed (Participants) | 791 | 805
  Change at Cycle 2: Systemic Therapy SE | 24.1 (18.1) | 18.3 (16.6)
  Change at Cycle 3: Systemic Therapy SE: number analyzed (Participants) | 793 | 812
  Change at Cycle 3: Systemic Therapy SE | 23.4 (17.8) | 15.1 (15.5)
  Change at Cycle 4: Systemic Therapy SE: number analyzed (Participants) | 793 | 814
  Change at Cycle 4: Systemic Therapy SE | 23.1 (18.1) | 13.2 (15.4)
  Change at Cycle 5: Systemic Therapy SE: number analyzed (Participants) | 793 | 806
  Change at Cycle 5: Systemic Therapy SE | 20.0 (17.6) | 11.8 (14.7)
  Change at Cycle 9: Systemic Therapy SE: number analyzed (Participants) | 772 | 770
  Change at Cycle 9: Systemic Therapy SE | 9.5 (13.1) | 10.4 (14.0)
  Change at Cycle 14: Systemic Therapy SE: number analyzed (Participants) | 755 | 730
  Change at Cycle 14: Systemic Therapy SE | 7.5 (12.9) | 9.8 (13.9)
  Change at EoT: Systemic Therapy SE: number analyzed (Participants) | 785 | 793
  Change at EoT: Systemic Therapy SE | 7.2 (13.4) | 8.5 (13.9)
  Change at FU Month 6: Systemic Therapy SE: number analyzed (Participants) | 745 | 726
  Change at FU Month 6: Systemic Therapy SE | 5.8 (12.3) | 4.2 (12.5)
  Change at FU Month 12: Systemic Therapy SE: number analyzed (Participants) | 716 | 705
  Change at FU Month 12: Systemic Therapy SE | 5.4 (12.9) | 4.2 (13.0)
  Change at FU Month 18: Systemic Therapy SE: number analyzed (Participants) | 0 | 0
  Baseline: Upset by Hair Loss Item: number analyzed (Participants) | 205 | 213
  Baseline: Upset by Hair Loss Item | 13.2 (23.7) | 14.2 (22.9)
  Change at Cycle 1: Upset by Hair Loss Item: number analyzed (Participants) | 169 | 168
  Change at Cycle 1: Upset by Hair Loss Item | 35.1 (37.3) | 25.2 (35.1)
  Change at Cycle 2: Upset by Hair Loss Item: number analyzed (Participants) | 152 | 130
  Change at Cycle 2: Upset by Hair Loss Item | 28.7 (36.0) | 21.8 (36.6)
  Change at Cycle 3: Upset by Hair Loss Item: number analyzed (Participants) | 132 | 98
  Change at Cycle 3: Upset by Hair Loss Item | 28.8 (36.3) | 21.4 (38.4)
  Change at Cycle 4: Upset by Hair Loss Item: number analyzed (Participants) | 136 | 83
  Change at Cycle 4: Upset by Hair Loss Item | 28.4 (37.1) | 19.7 (34.2)
  Change at Cycle 5: Upset by Hair Loss Item: number analyzed (Participants) | 130 | 83
  Change at Cycle 5: Upset by Hair Loss Item | 26.4 (36.8) | 10.0 (36.3)
  Change at Cycle 9: Upset by Hair Loss Item: number analyzed (Participants) | 85 | 72
  Change at Cycle 9: Upset by Hair Loss Item | 11.8 (33.6) | 6.0 (36.8)
  Change at Cycle 14: Upset by Hair Loss Item: number analyzed (Participants) | 68 | 53
  Change at Cycle 14: Upset by Hair Loss Item | 9.3 (32.5) | 2.5 (26.0)
  Change at EoT: Upset by Hair Loss Item: number analyzed (Participants) | 75 | 63
  Change at EoT: Upset by Hair Loss Item | 17.3 (33.9) | 0.0 (28.1)
  Change at FU Month 6: Upset by Hair Loss Item: number analyzed (Participants) | 86 | 67
  Change at FU Month 6: Upset by Hair Loss Item | 6.2 (26.8) | -3.5 (21.0)
  Change at FU Month 12: Upset by Hair Loss Item: number analyzed (Participants) | 84 | 71
  Change at FU Month 12: Upset by Hair Loss Item | 2.4 (28.7) | -2.8 (29.7)
  Change at FU Month 18: Upset by Hair Loss Item: number analyzed (Participants) | 0 | 0
  Baseline: Body Image: number analyzed (Participants) | 841 | 867
  Baseline: Body Image | 78.5 (23.2) | 78.9 (24.2)
  Change at Cycle 1: Body Image: number analyzed (Participants) | 808 | 834
  Change at Cycle 1: Body Image | -13.7 (23.5) | -13.3 (23.1)
  Change at Cycle 2: Body Image: number analyzed (Participants) | 788 | 801
  Change at Cycle 2: Body Image | -12.7 (23.9) | -10.1 (23.9)
  Change at Cycle 3: Body Image: number analyzed (Participants) | 787 | 807
  Change at Cycle 3: Body Image | -11.5 (24.8) | -6.6 (22.6)
  Change at Cycle 4: Body Image: number analyzed (Participants) | 788 | 810
  Change at Cycle 4: Body Image | -11.4 (24.8) | -5.9 (23.2)
  Change at Cycle 5: Body Image: number analyzed (Participants) | 790 | 802
  Change at Cycle 5: Body Image | -10.5 (24.6) | -5.0 (22.6)
  Change at Cycle 9: Body Image: number analyzed (Participants) | 768 | 766
  Change at Cycle 9: Body Image | -5.9 (22.8) | -4.2 (21.7)
  Change at Cycle 14: Body Image: number analyzed (Participants) | 750 | 726
  Change at Cycle 14: Body Image | -4.5 (23.6) | -2.4 (23.2)
  Change at EoT: Body Image: number analyzed (Participants) | 783 | 785
  Change at EoT: Body Image | -3.3 (23.1) | -2.9 (22.8)
  Change at FU Month 6: Body Image: number analyzed (Participants) | 740 | 720
  Change at FU Month 6: Body Image | -1.3 (23.4) | 0.3 (23.3)
  Change at FU Month 12: Body Image: number analyzed (Participants) | 712 | 703
  Change at FU Month 12: Body Image | 0.0 (24.2) | 0.7 (23.5)
  Change at FU Month 18: Body Image: number analyzed (Participants) | 0 | 0
  Baseline: Future Perspectives (FP): number analyzed (Participants) | 842 | 868
  Baseline: Future Perspectives (FP) | 49.3 (31.4) | 49.8 (30.9)
  Change at Cycle 1: FP: number analyzed (Participants) | 805 | 836
  Change at Cycle 1: FP | -1.3 (30.3) | -0.3 (31.1)
  Change at Cycle 2: FP: number analyzed (Participants) | 786 | 803
  Change at Cycle 2: FP | 1.4 (31.7) | 3.7 (30.4)
  Change at Cycle 3: FP: number analyzed (Participants) | 786 | 811
  Change at Cycle 3: FP | 3.2 (32.0) | 6.5 (30.1)
  Change at Cycle 4: FP: number analyzed (Participants) | 787 | 814
  Change at Cycle 4: FP | 4.2 (31.7) | 7.8 (30.5)
  Change at Cycle 5: FP: number analyzed (Participants) | 787 | 804
  Change at Cycle 5: FP | 5.9 (32.4) | 9.7 (30.7)
  Change at Cycle 9: FP: number analyzed (Participants) | 762 | 767
  Change at Cycle 9: FP | 8.2 (32.2) | 8.4 (31.3)
  Change at Cycle 14: FP: number analyzed (Participants) | 752 | 726
  Change at Cycle 14: FP | 9.5 (32.0) | 7.9 (33.4)
  Change at EoT: FP: number analyzed (Participants) | 782 | 787
  Change at EoT: FP | 8.5 (32.6) | 7.6 (32.3)
  Change at FU Month 6: FP: number analyzed (Participants) | 740 | 720
  Change at FU Month 6: FP | 10.5 (31.3) | 12.6 (32.6)
  Change at FU Month 12: FP: number analyzed (Participants) | 711 | 703
  Change at FU Month 12: FP | 15.0 (34.0) | 13.1 (33.2)
  Change at FU Month 18: FP: number analyzed (Participants) | 0 | 0
  Baseline: Sexual Enjoyment: number analyzed (Participants) | 369 | 380
  Baseline: Sexual Enjoyment | 43.4 (32.1) | 46.7 (34.8)
  Change at Cycle 1: Sexual Enjoyment: number analyzed (Participants) | 233 | 260
  Change at Cycle 1: Sexual Enjoyment | -5.9 (26.8) | -8.2 (27.0)
  Change at Cycle 2: Sexual Enjoyment: number analyzed (Participants) | 196 | 227
  Change at Cycle 2: Sexual Enjoyment | -9.5 (30.2) | -10.7 (29.2)
  Change at Cycle 3: Sexual Enjoyment: number analyzed (Participants) | 205 | 235
  Change at Cycle 3: Sexual Enjoyment | -11.4 (26.8) | -8.9 (31.6)
  Change at Cycle 4: Sexual Enjoyment: number analyzed (Participants) | 190 | 228
  Change at Cycle 4: Sexual Enjoyment | -11.9 (30.6) | -9.2 (28.3)
  Change at Cycle 5: Sexual Enjoyment: number analyzed (Participants) | 204 | 224
  Change at Cycle 5: Sexual Enjoyment | -14.2 (28.1) | -8.8 (30.4)
  Change at Cycle 9: Sexual Enjoyment: number analyzed (Participants) | 221 | 220
  Change at Cycle 9: Sexual Enjoyment | -9.4 (29.5) | -7.4 (30.9)
  Change at Cycle 14: Sexual Enjoyment: number analyzed (Participants) | 203 | 213
  Change at Cycle 14: Sexual Enjoyment | -3.9 (28.6) | -9.7 (31.4)
  Change at EoT: Sexual Enjoyment: number analyzed (Participants) | 224 | 236
  Change at EoT: Sexual Enjoyment | -6.5 (29.2) | -9.7 (29.4)
  Change at FU Month 6: Sexual Enjoyment: number analyzed (Participants) | 212 | 223
  Change at FU Month 6: Sexual Enjoyment | -4.6 (28.8) | -3.0 (30.5)
  Change at FU Month 12: Sexual Enjoyment: number analyzed (Participants) | 212 | 204
  Change at FU Month 12: Sexual Enjoyment | -5.7 (30.9) | -2.3 (31.0)
  Change at FU Month 18: Sexual Enjoyment: number analyzed (Participants) | 0 | 0
  Baseline: Sexual Function: number analyzed (Participants) | 819 | 829
  Baseline: Sexual Function | 16.7 (22.3) | 18.3 (22.9)
  Change at Cycle 1: Sexual Function: number analyzed (Participants) | 757 | 779
  Change at Cycle 1: Sexual Function | -2.3 (18.9) | -3.5 (18.4)
  Change at Cycle 2: Sexual Function: number analyzed (Participants) | 728 | 745
  Change at Cycle 2: Sexual Function | -4.8 (19.9) | -4.4 (18.4)
  Change at Cycle 3: Sexual Function: number analyzed (Participants) | 734 | 740
  Change at Cycle 3: Sexual Function | -5.6 (19.6) | -3.3 (19.0)
  Change at Cycle 4: Sexual Function: number analyzed (Participants) | 726 | 743
  Change at Cycle 4: Sexual Function | -6.8 (19.7) | -3.4 (17.9)
  Change at Cycle 5: Sexual Function: number analyzed (Participants) | 730 | 738
  Change at Cycle 5: Sexual Function | -5.9 (19.5) | -3.0 (19.5)
  Change at Cycle 9: Sexual Function: number analyzed (Participants) | 710 | 704
  Change at Cycle 9: Sexual Function | -3.4 (19.3) | -1.8 (20.8)
  Change at Cycle 14: Sexual Function: number analyzed (Participants) | 696 | 671
  Change at Cycle 14: Sexual Function | -1.8 (20.0) | -2.8 (20.6)
  Change at EoT: Sexual Function: number analyzed (Participants) | 716 | 724
  Change at EoT: Sexual Function | -1.5 (20.9) | -1.7 (19.7)
  Change at FU Month 6: Sexual Function: number analyzed (Participants) | 675 | 658
  Change at FU Month 6: Sexual Function | 1.6 (22.6) | 0.6 (20.4)
  Change at FU Month 12: Sexual Function: number analyzed (Participants) | 651 | 639
  Change at FU Month 12: Sexual Function | 0.9 (21.7) | 0.9 (20.9)
  Change at FU Month 18: Sexual Function: number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Clinically Meaningful Deterioration in the Global Health Status/ Quality of Life and Functional (Physical, Role, and Cognitive) Subscales of the QLQ-C30 From First HER2-Targeted Treatment
Description: The time to clinically meaningful deterioration in the global health status/Quality of life and Functional (Physical, Role, and Cognitive) subscales of the the QLQ-C30 was assessed from the time of the HER2-Targeted treatment to the worsening in the respective scales. Clinically meaningful deterioration is defined as a decrease in score of 10 points in Physical functioning and HRQoL; decrease of 7 points in Cognitive functioning, and decrease of 14 points in Role functioning.
Time Frame: From start of HER-2 targeted treatment up to 18 months after treatment discontinuation. The median time to clinically meaningful deterioration was assessed based on the data collection described above.
Population: The Patient Reported Outcome (PRO) Population includes participants with both a baseline assessment and at least one post-baseline assessment in any PRO items. This subset population includes only participants who received HER2-targeted therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
Number analyzed (Participants) | 864 | 884
months
  GHS/QoL Score: number analyzed (Participants) | 858 | 879
  GHS/QoL Score | 2.73 [2.10 to 2.83] | 13.57 [9.20 to 21.91]
  Physical Function: number analyzed (Participants) | 861 | 879
  Physical Function | 25.53 [13.34 to NA] — Upper limit not reached. | NA [27.43 to NA] — The median and upper limit were not reached.
  Role Function: number analyzed (Participants) | 859 | 880
  Role Function | 2.23 [2.10 to 2.79] | 9.92 [9.00 to 14.36]
  Cognitive Function: number analyzed (Participants) | 858 | 879
  Cognitive Function | 5.49 [2.79 to 5.82] | 9.46 [8.57 to 12.91]

ADVERSE EVENTS:
Time Frame: From randomization to approximately 7.5 years
Description: AEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0. 8 participants were randomized but did not receive any study treatment (5 in the AC-THP arm, 3 in the AC-KP arm). 16 participants in the AC-THP, and 13 in the AC-KP arm only received AC but no HER2 targeted therapy and were consequently assigned to the AC-THP arm for safety analysis.
Arm/Group | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab
All-Cause Mortality (participants affected / at risk) | 45/926 | 55/912
Serious Adverse Events (participants affected / at risk) | 216/926 | 195/912
Other Adverse Events (participants affected / at risk) | 902/926 | 902/912
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane (N=926) | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab (N=912)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 51 (55) | 31 (32)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 16 (18) | 10 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 5 (5) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 4 (4)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 20 (22) | 8 (8)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10) | 7 (7)
Catheter site pain (General disorders) | 0 (0) | 1 (3)
Catheter site vesicles (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 13 (14) | 19 (22)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 0 (0) | 3 (3)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 4 (4)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 2 (3)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Incision site abscess (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Mastitis (Infections and infestations) | 8 (9) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 7 (8) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 12 (12) | 12 (12)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (2)
Postoperative wound infection (Infections and infestations) | 2 (3) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 8 (8)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 9 (9)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine increased (Investigations) | 1 (1) | 0 (0)
Blood pressure decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram repolarisation abnormality (Investigations) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 3 (3) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 2 (2)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anthracycline Followed by Trastuzumab, Pertuzumab, and Taxane (N=926) | Anthracycline Followed by Trastuzumab Emtansine and Pertuzumab (N=912)
Anaemia (Blood and lymphatic system disorders) | 184 (249) | 174 (243)
Leukopenia (Blood and lymphatic system disorders) | 73 (134) | 51 (96)
Neutropenia (Blood and lymphatic system disorders) | 232 (411) | 220 (403)
Thrombocytopenia (Blood and lymphatic system disorders) | 25 (29) | 162 (297)
Dry eye (Eye disorders) | 62 (69) | 75 (87)
Lacrimation increased (Eye disorders) | 112 (120) | 73 (75)
Vision blurred (Eye disorders) | 42 (44) | 46 (49)
Abdominal pain (Gastrointestinal disorders) | 83 (103) | 86 (110)
Abdominal pain upper (Gastrointestinal disorders) | 83 (90) | 87 (110)
Constipation (Gastrointestinal disorders) | 287 (369) | 299 (413)
Diarrhoea (Gastrointestinal disorders) | 605 (1158) | 405 (759)
Dry mouth (Gastrointestinal disorders) | 63 (68) | 105 (116)
Dyspepsia (Gastrointestinal disorders) | 123 (146) | 106 (123)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 58 (64) | 39 (41)
Gingival bleeding (Gastrointestinal disorders) | 6 (6) | 57 (64)
Haemorrhoids (Gastrointestinal disorders) | 58 (71) | 46 (50)
Nausea (Gastrointestinal disorders) | 596 (1034) | 605 (1246)
Stomatitis (Gastrointestinal disorders) | 276 (441) | 228 (338)
Vomiting (Gastrointestinal disorders) | 243 (358) | 289 (502)
Asthenia (General disorders) | 121 (222) | 131 (254)
Chills (General disorders) | 40 (45) | 67 (79)
Fatigue (General disorders) | 439 (672) | 419 (659)
Influenza like illness (General disorders) | 26 (33) | 62 (72)
Malaise (General disorders) | 42 (58) | 60 (90)
Mucosal inflammation (General disorders) | 156 (213) | 111 (134)
Oedema peripheral (General disorders) | 156 (173) | 74 (91)
Pyrexia (General disorders) | 175 (242) | 227 (353)
Conjunctivitis (Infections and infestations) | 49 (51) | 42 (44)
Nasopharyngitis (Infections and infestations) | 175 (269) | 171 (257)
Paronychia (Infections and infestations) | 53 (59) | 50 (54)
Upper respiratory tract infection (Infections and infestations) | 139 (197) | 125 (176)
Urinary tract infection (Infections and infestations) | 73 (99) | 63 (82)
Infusion related reaction (Injury, poisoning and procedural complications) | 115 (132) | 126 (157)
Radiation skin injury (Injury, poisoning and procedural complications) | 207 (210) | 205 (213)
Alanine aminotransferase increased (Investigations) | 108 (134) | 301 (418)
Aspartate aminotransferase increased (Investigations) | 98 (113) | 317 (431)
Blood alkaline phosphatase increased (Investigations) | 20 (24) | 85 (100)
Blood bilirubin increased (Investigations) | 4 (6) | 80 (127)
Ejection fraction decreased (Investigations) | 61 (72) | 29 (35)
Neutrophil count decreased (Investigations) | 83 (148) | 75 (135)
Platelet count decreased (Investigations) | 15 (21) | 143 (203)
Weight decreased (Investigations) | 57 (61) | 79 (82)
Decreased appetite (Metabolism and nutrition disorders) | 241 (348) | 244 (371)
Hypokalaemia (Metabolism and nutrition disorders) | 41 (50) | 67 (102)
Arthralgia (Musculoskeletal and connective tissue disorders) | 289 (397) | 261 (338)
Back pain (Musculoskeletal and connective tissue disorders) | 120 (138) | 93 (111)
Bone pain (Musculoskeletal and connective tissue disorders) | 70 (94) | 58 (71)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 86 (92) | 97 (129)
Myalgia (Musculoskeletal and connective tissue disorders) | 214 (255) | 152 (195)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 119 (154) | 114 (136)
Dizziness (Nervous system disorders) | 117 (140) | 105 (138)
Dysgeusia (Nervous system disorders) | 180 (205) | 162 (177)
Headache (Nervous system disorders) | 234 (328) | 261 (419)
Neuropathy peripheral (Nervous system disorders) | 163 (204) | 140 (164)
Paraesthesia (Nervous system disorders) | 85 (102) | 101 (129)
Peripheral sensory neuropathy (Nervous system disorders) | 214 (236) | 193 (209)
Taste disorder (Nervous system disorders) | 56 (67) | 60 (69)
Anxiety (Psychiatric disorders) | 58 (63) | 42 (48)
Depression (Psychiatric disorders) | 52 (54) | 52 (54)
Insomnia (Psychiatric disorders) | 171 (204) | 155 (190)
Breast pain (Reproductive system and breast disorders) | 45 (57) | 55 (65)
Cough (Respiratory, thoracic and mediastinal disorders) | 148 (189) | 157 (190)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 (87) | 79 (91)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 182 (226) | 333 (487)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 111 (132) | 100 (123)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 77 (87) | 82 (96)
Alopecia (Skin and subcutaneous tissue disorders) | 629 (651) | 598 (616)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 52 (59) | 53 (60)
Dry skin (Skin and subcutaneous tissue disorders) | 132 (143) | 100 (112)
Erythema (Skin and subcutaneous tissue disorders) | 86 (100) | 75 (82)
Nail discolouration (Skin and subcutaneous tissue disorders) | 104 (104) | 76 (78)
Nail disorder (Skin and subcutaneous tissue disorders) | 68 (72) | 43 (43)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 66 (74) | 25 (31)
Pruritus (Skin and subcutaneous tissue disorders) | 169 (222) | 126 (151)
Rash (Skin and subcutaneous tissue disorders) | 249 (353) | 214 (290)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 47 (56) | 42 (59)
Hot flush (Vascular disorders) | 167 (190) | 100 (110)
Hypertension (Vascular disorders) | 36 (51) | 63 (83)
Lymphoedema (Vascular disorders) | 68 (70) | 30 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2015-07-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT01966471/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT01966471/SAP_001.pdf